CLINICAL TRIAL: NCT03851640
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled Phase III Clinical Trial Evaluating the Efficacy and Safety of HC-1119 Soft Capsules in Patients with Metastatic Castration-Resistant Prostate Cancer (mCRPC) Who Have Failed Treatments with Abiraterone Acetate and Docetaxel.
Brief Title: A Trial Evaluating the Efficacy and Safety of HC-1119 Soft Capsules in Patients with Metastatic Castration-Resistant Prostate Cancer (mCRPC).
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hinova Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: HC-1119-04
Record Dates: First submitted 2019-02-17; First posted 2019-02-22 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2024-11

CONDITIONS: MCRPC
MeSH Terms: interventions — enzalutamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HC-1119 (Experimental): 80mg;
  Interventions: Drug: HC-1119
- placebo (Placebo Comparator): 80mg;
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: HC-1119 — oral
  Arms: HC-1119
Drug: placebo — oral
  Arms: placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, Phase 3 clinical study evaluating the efficacy and safety of HC-1119 soft capsules versus placebo in mCRPC patients who have failed or become intolerant to the treatments with both abiraterone acetate and docetaxel, or who are not suitable for docetaxel treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Males aged ≥18 years at screening and voluntary to participate in the study and sign the informed consent form.
2. Subjects with histologically or cytologically confirmed prostate adenocarcinoma, with no small cell features.
3. In the case of medical or surgical castration, during or after the last treatment before screening, there are signs of progressive disease determined according to the PCWG3 criteria, defined as satisfying one or more of the following 3 criteria:

   1. PSA progression; at least 2 episodes of increased PSA levels that are measured ≥1 week apart; PSA ≥ 1 μg/L (1 ng/mL) in the screening period;
   2. Progression of soft tissue lesions as defined by RECIST 1.1;
   3. The progression of bone lesions is defined as at least two new lesions discovered by bone scan; ambiguous results can be confirmed using another imaging technique (e.g., CT or MRI).
4. Metastatic diseases confirmed by imaging examinations during the screening period (the status of metastasis refers to the presence of metastatic lesions confirmed by bone scan and/or CT/MRI scan).
5. For patients who have undergone orchiectomy or are being treated by medical castration therapy, their androgen blockade therapy is maintained by luteinizing hormone-releasing hormone agonists or antagonists during the study period (including the follow-up period), and their serum testosterone levels are ≤ 1.73 nmol/L (50 ng/dL) during screening visits.
6. Patients who have failed previous treatments of prostate cancer with abiraterone acetate or who are intolerant to treatments with abiraterone acetate.
7. Patients who have failed previous chemotherapy of prostate cancer with docetaxel or who are intolerant to treatments with docetaxel, or who are not suitable for docetaxel treatment during screening. Patients who are not suitable for docetaxel treatment during screening and do not plan to use cytotoxic chemotherapy within 6 months after the informed discussion are eligible.
8. Expected survival of ≥ 3 months.
9. ECOG performance status score of 0-2.
10. Laboratory tests must meet the following criteria:

    1. Blood routine examination: Hemoglobin (Hb) ≥ 85 g/L; white blood cell (WBC) ≥ 3.0 x 109/L; platelet (PLT) ≥ 75 x 109/L;
    2. Liver function: Total bilirubin (TBIL) ≤ 1.5 x ULN; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN (for patients without liver metastasis) or ≤ 5 x ULN (for patients with liver metastasis); albumin (ALB) ≥ 25 g/L;
    3. Renal function: serum creatinine (SCr) ≤ 1.5 x ULN.
11. Willing to use reliable contraceptive measures (such as condoms) and not to donate sperms throughout the study period and within 3 months after the last dose.

Exclusion Criteria:

Subjects with any of the following conditions should not be enrolled:

1. Received any anti-prostate cancer treatment within 4 weeks before randomization, including chemotherapy, immunotherapy, targeted therapy, estrogen therapy, anti-androgen therapy, systemic radiotherapy, treatments with traditional Chinese medicines for anticancer, or treatments with interventional drugs of other clinical trials; palliative radiotherapy or surgery for bone metastatic or soft tissue lesions should be completed >14 days prior to baseline imaging examinations; the lesions treated by palliative radiotherapy should not be the targeted lesions of subsequent RECIST 1.1 assessment. Androgen blockade therapy that is maintained by a luteinizing hormone releasing hormone agonist or antagonist.
2. Previously received any of novel androgen receptor inhibitors (e.g., Enzalutamide, Apalutamide, Darolutamide, SHR3680, Proxalutamide, or HC-1119).
3. Patients with brain or central nervous system metastases are known (if a brain or central nervous system metastasis is suspected, a CT/MRI scan of the head is required)
4. Patients with known serious cardiovascular diseases, including any of the following:

   1. A myocardial infarction or thrombotic event occurred in the past 6 months;
   2. Known unstable angina;
   3. Heart failure of Grade III or IV according to the New York Heart Association (NYHA) criteria;
   4. QT interval of > 500 ms during screening visits;
   5. Resting systolic blood pressure of >170 mmHg or diastolic blood pressure of >105 mmHg suggesting uncontrolled hypertension during screening visits.
5. The toxicity of previous treatment has not been eliminated before the start of the study treatment; toxic reaction of grade 2 or above (except for hair loss) according to the CTCAE 5.0 grading scale remains.
6. Clinically significant gastrointestinal abnormalities that may affect the intake, transport or absorption of drugs (for example, inability to swallow, chronic diarrhea or intestinal obstruction, and patients had total gastrectomy).
7. Patients with a history of serious diseases in the central nervous system. Patients with a history of epilepsy or any history of diseases that may induce epilepsy, including unexplained loss of consciousness or transient ischemic attack.
8. Patients who have been diagnosed in the past 5 years with other malignant tumors in addition to prostate cancer, except patients with cured basal or squamous cell skin cancer and superficial bladder tumors (Ta, Tis, and T1).
9. Patients with a history of allogeneic bone marrow or organ transplantation who require continued medical treatment.
10. Patients with known congenital or acquired immunodeficiency, active hepatitis, active tuberculosis or other active infections.
11. Patients known to be allergic to androgen receptor inhibitors.
12. The investigator believes that the patients are unfit for this study (e.g., the treatments will not benefit the patients the most, inadequate patient compliance, etc.).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 417 (Estimated)
Dates: Start 2019-04-12 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Radiographic Progression-Free Survival (rPFS) | From signing informed consent up to approximately 30 months

SECONDARY OUTCOMES:
Overall Survival (OS) | From signing informed consent up to approximately 30 months
Time to progression (TTP) | From signing informed consent up to approximately 30 months
Objective response rate (ORR) | From signing informed consent up to approximately 30 months
Disease control rate (DCR) | From signing informed consent up to approximately 30 months
Response rate of prostate specific antigen (PSA) | From signing informed consent up to approximately 30 months
Time to prostate specific antigen(PSA) progression (TTPP) | From signing informed consent up to approximately 30 months
Number of patients with adverse events | From signing informed consent up to approximately 30 months
  Safety measures

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No